CLINICAL TRIAL: NCT00420810
Title: A Double-Blind, Placebo Controlled, Randomized, Cross-Over Polysomnographic Study of MK0928 15 mg in Adult Patients With Primary Insomnia
Brief Title: Adult Polysomnography Primary Insomnia Cross Over Study (0928-049)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-049; 2006_514
Record Dates: First submitted 2007-01-05; First posted 2007-01-11 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Duration of Therapy

INTERVENTIONS:
Drug: MK0928 / Duration of Treatment : 8 Weeks

SUMMARY:
The purpose of this study is determine whether this drug will improve your insomnia in terms of decreasing your time to fall asleep and allowing you to stay asleep longer. The drug will be compared against placebo in order to determine if there's a difference.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Insomnia
* Patient is willing to stay overnight at a sleep laboratory for a total of 7 nights
* Patient is willing to avoid alcohol on PSG visits
* Patient will avoid napping during the course of the study
* Patient's bedtime is between 9pm and 1am

Exclusion Criteria:

* History of substance abuse, bipolar disorder or psychotic disorder
* Difficulty sleeping due to other medical condition
* History of narcolepsy, circadian rhythm sleep disorder, parasomnia, sleep apnea, periodic limb movements or restless legs syndrome
* History of neoplastic malignancy within the last 5 years
* Positive alcohol breath test during the screening visits

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138
Dates: Start 2006-09; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Wake after sleep onset and Latency to persistent sleep

SECONDARY OUTCOMES:
Subjective total sleep time and subjective time to sleep onset

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC